CLINICAL TRIAL: NCT00638807
Title: A Double-Blind, Placebo Controlled Study of the Efficacy and Tolerability of Once Daily Celebrex (Celecoxib) vs. Placebo in the Treatment of Subjects With Osteoarthritis of the Knee Non-Responsive to Naproxen and Ibuprofen
Brief Title: Safety and Efficacy of Celecoxib Versus Placebo in the Treatment of Knee Osteoarthritis in Patients Who Were Unresponsive to Naproxen and Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191082
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Celecoxib — 200 mg oral capsule once daily with morning meal for 6 weeks
  Arms: A
Other: Placebo — Matched oral placebo for 6 weeks
  Arms: B

SUMMARY:
To compare the efficacy and safety of celecoxib versus placebo for the treatment of knee osteoarthritis (OA) in patients who were unresponsive to prescription strength naproxen and ibuprofen or who could not tolerate prescription strength naproxen and ibuprofen

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Diagnosed, active, and symptomatic OA of the knee in a flare state with a functional capacity class of I-III at baseline visit
* Failed adequate trials of both naproxen and ibuprofen (prescription strength) within the past 5 years due to lack of efficacy, tolerability, or both; duration of prescription strength ibuprofen and naproxen must have been a minimum of 2 weeks for each drug at the respective recommended doses if failure was due to lack of efficacy, and for any duration if failure was due to lack of tolerability

Exclusion Criteria:

Exclusion criteria:

* Inflammatory arthritis or gout/pseudo-gout with acute flare within the past 2 years (subjects with fibrositis or fibromyalgia will not be excluded)
* Received acetaminophen within 24 hours of the baseline visit
* Use of a mobility assisting device for less than six weeks prior to study screening or use of a walker
* History of gastrointestinal (GI) perforation, obstruction, or bleeding
* Diagnosed or treated for GI ulcer within 60 days prior to first dose of study medication
* Received corticosteroids or hyaluronic acid within certain timeframe before study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2003-12; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Patient's Assessment of Arthritis Pain, according to visual analog scale (VAS) | Week 6

SECONDARY OUTCOMES:
Patient's Assessment of Arthritis Pain, according to VAS | Week 2
The Western Ontario and McMaster Universities Osteoarthritis Index | Week 6
Patient's and Physician's Global Assessment of Arthritis | Weeks 2 and 6
The Medical Outcomes Study Sleep Scale | Week 6
Adverse events | Weeks 0-6
Laboratory tests | Week 6
Vital signs | Week 6
Physical examination | Week 6
Serious adverse events | Up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (31):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Buena Park, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Bozeman, Montana
  - Pfizer Investigational Site, Trenton, New Jersey
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191082&StudyName=Safety%20and%20Efficacy%20of%20Celecoxib%20Versus%20Placebo%20in%20the%20Treatment%20of%20Knee%20Osteoarthritis%20in%20Patients%20who%20were%20Unresponsive%20to%20Naproxen%20